CLINICAL TRIAL: NCT02434679
Title: Dynamic of the Acquisition of Antibiotic Resistance in Integrons in Neonatology Newborns
Acronym: DAIR3N
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I13024 DAIR3N
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Bacteriology
Keywords: antibiotics resistance integrons; neonatology newborns; digestive acquisition; dynamic of the acquisition of integrons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The meconium or the first stool will be sampled at D0. The stool will then be sampled: at D7, at D21 and every 15 days until the day of discharge.
  If the NB has no stool on the given day, a period of 3 more days will be accepted from the day the sampling was planned. After this period, "no sample" will be stated.
  Meconiums and stool must be sampled in sterile jars, labelled and sent with the designation "DAIR3N protocol" to the bacteriology laboratory of each center. If the local laboratory cannot seed the samples 7 days a week, stool samples can be kept maximum 48h at +4°C before management.
  In the mother
  Vaginal sample will be taken during the delivery according to care practices of each center if:
  it is a preterm vaginal delivery, early membrane rupture happens, there is a threat of very preterm delivery. About 55% of inclusions should be subject to this type of sampling. Sampling of mother's stool will be asked at the inclusion.
Oversight: Data Monitoring Committee: No

SUMMARY:
Antibiotic resistance is a major public health issue as multiresistant bacteria (MRB) are increasing. Among the actions to control resistance, one is an interesting lead: to prevent the emergence of resistant bacteria by limiting possibilities for bacteria to acquire resistance. Mechanisms of resistance genes acquisition are deeply studied but there are few data on the dynamic of acquisition over time. Among the genetic components that disseminate resistance genes, resistance integrons (RI) play a major role in the acquisition and dissemination of antibiotic resistance in gram-negative bacteria. The digestive tract of the newborn (NB), which is initially sterile, is colonized by a bacterial microbiota during the first days of life. It thus appears to be an appropriate model to study the dynamic of resistance acquisition. This project intends to follow the NB of neonatology over time in order to study the dynamic of the digestive acquisition of RI and MRB

ELIGIBILITY:
Inclusion Criteria:

* Mother-child pairs that will be included in the study will be the pairs of all the NB, born in the center (in born) and hospitalized in the neonatology units of each center:

with a predictable stay ≥ 3 weeks in the unit

Exclusion Criteria:

NB will not be included if:

* They exhibit a birth defect, especially on the digestive tract
* They are secondarily hospitalized after a postnatal transfer (out born).
* The parents express their objection for the child to take part in the study
* The stool sample of the mother has not been received

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mother-child pairs of all the NB, born in the center and hospitalized in the neonatology units of each center with a predictable stay ≥ 3 weeks in the unit
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The occurrence over time of digestive acquisition of any type of RI | 3 weeks

SECONDARY OUTCOMES:
The occurrence over time of digestive acquisition of severals type of RI | 3 weeks
  "intI1" whenever the gene encoding a class 1 integrase will be detected "intI2" whenever the gene encoding a class 2 integrase will be detected "intI3" whenever the gene encoding a class 3 integrase will be detected An association: "intI1+intI2", "intI1+intI3", "intI2+intI3", "intI1+intI2+intI3" will also be searched.
Occurrence over time of digestive acquisition of MRB in NB hospitalized in neonatology units | 3 weeks
  Occurrence over time of digestive acquisition of MRB in NB hospitalized in neonatology units

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BEDU, MD, Principal Investigator — University Hospital, Limoges
Locations (5):
- France (5):
  - Hospital center, Bayonne
  - University Hospital, Bordeaux
  - University hospital, Limoges
  - Hospital center, Pau
  - University Hospital, Toulouse